CLINICAL TRIAL: NCT05410431
Title: Atypical Intraorbital Dermoid and Epidermoid Cyst: A Single Institution Cross-sectional Retrospective Study
Brief Title: Intraorbital Dermoid/Epidermoid Cyst
Status: Completed | Type: Observational
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohsen Pourazizi, Principal Investigator, Isfahan University of Medical Sciences
Other Study IDs: IR.MUI.MED.REC.1399.1052
Record Dates: First submitted 2022-05-31; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Dermoid Cyst of Orbit

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical and radiologic manifestations of rare presentations of Dermoid cyst

SUMMARY:
Intraorbital epidermoid and dermoid cyst (DC) has been reported in the literature rarely. The current study evaluates clinicopathologic, radiologic, and management of intraorbital DC cases over ten years.

ELIGIBILITY:
Inclusion Criteria:

* Those who had an excision biopsy with histology indicative of dermoid/epidermoid cyst

Exclusion Criteria:

* Other cystic lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Intraorbital Dermoid and Epidermoid Cyst
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Histopathology report | Ten years
  cyst pathology
Magnetic Resonance Imaging report | Ten years
  The cyst features
Surgery technique | Ten years
  Managing the cyst

IPD SHARING:
Plan to Share IPD: Undecided